CLINICAL TRIAL: NCT01029821
Title: Low-Molecular-Weight Heparin for DVT Prophylaxis After Open Reduction and Internal Fixation of Ankle Fractures: A Randomized, Prospective Trial
Brief Title: Low-Molecular-Weight Heparin (LMWH) for Deep Venous Thrombosis (DVT) Prophylaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Elaine Pugh, UTennessee
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pugh-2
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Deep Venous Thrombosis
Keywords: Low-Molecular-Weight-Heparin; Open Reduction and Internal Fixation; Thromboprophylaxis
MeSH Terms: conditions — Venous Thrombosis | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-Molecular-Weight Heparin for DVT (Other): Low-Molecular-Weight Heparin for DVT Prophylaxis after Open Reduction and Internal Fixation of ankle fractures
  Interventions: Drug: Low-Molecular-Weight Heparin

INTERVENTIONS:
Drug: Low-Molecular-Weight Heparin — Isolated Ankle Fracture Single planned operation

SUMMARY:
1. The use of LMWH following open reduction and internal fixation of ankle fractures will reduce the number of thrombi formed.
2. The rates of clinically significant DVT will be equivalent between two groups.

DETAILED DESCRIPTION:
Routine use of thromboprophylaxis may be over treatment and definitely increases healthcare costs. While prophylaxis may reduce the number of thrombi formed the exact number and clinical significance of these is unknown. This study seeks to answer the question of whether or not DVT prophylaxis with low-molecular-weight heparin (LMWH) following ORIF of ankle fractures is warranted.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Surgical ankle fracture able to be definitively treated with one operation

Exclusion Criteria:

* Younger than 18 years of age
* Other significant injury
* Known hypercoagulable state
* History of bleeding disorder
* History of DVT

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
We will compare the rates of thrombi formation between the two groups. We will record any clinical significant thrombi or complications that arise from thrombi. We will record any complications related to administration of LMWH. | first post-operative office visit (usually 10-14 days)

SECONDARY OUTCOMES:
We may find that there is in fact significant benefit to giving prophylaxis to this subset of patients in the form of decreased rates of throb\mbus formation and the complications related to thrombi. The risk/benefit ratio should be favorable. | first post-operative office visit (10-14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Ingram, M.D., Principal Investigator — University of Tennessee
Locations (1):
- Erlanger Medical Center, Chattanooga, Tennessee, United States